CLINICAL TRIAL: NCT06100133
Title: Treat Autosomal Dominant Polycystic Kidney Disease With Oral Ketone Ester?
Acronym: ADKETONE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEFADPKD1
Record Dates: First submitted 2023-09-29; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: ADPKD
Keywords: ketone ester
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Repeated measures design to register the changes before and after treatment. Non-randomized, non-blinded, multi center prospective interventional cohort trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketone Ester (Experimental): Up to 100g ketone ester daily for 56 days
  Interventions: Dietary Supplement: Ketone ester

INTERVENTIONS:
Dietary Supplement: Ketone ester — Up to 100g ketone ester daily for 56 days
  Other Names: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (Ketone Ester)

SUMMARY:
The investigators are running a study to see if a special drink, called a "ketone ester", can help people with a type of kidney disease named "Autosomal Dominant Polycystic Kidney Disease" or ADPKD for short.

The investigators want to find out:

If it's easy for patients to take this drink every day for about 2 months. If it's safe and doesn't cause any problems. If it makes a difference in the size and function of the kidneys.

Who can join?

People between 16 to 70 years old who have ADPKD. Those with a certain amount of kidney size and function. People who haven't been on specific diets or lost a lot of weight recently. Women who are not breastfeeding and are using birth control. People with a body weight that is not too low or too high.

Who cannot join?

People who've been on a high-fat diet or skipped meals for a while recently. Those with other health conditions like diabetes or certain metabolic issues. Anyone who has a problem with getting an MRI scan. If participants are in another medical study right now.

The study will happen in two Belgian hospitals and is supported by the UZ Brussel's nephrology department. The investigators hope to include 20 people and start in November 2023.

ELIGIBILITY:
Inclusion Criteria:

* - ADPKD patients (diagnosis based on genetics or imaging) ≥ 16 and ≤ 70 years.
* Total Kidney Volume ≥ 600 mL.
* eGFR (CKD-EPI) ≥ 30 ml/min/1.73m2.
* Normal blood glucose, HbA1C and ketones.
* Women of childbearing potential who are non-lactating and using an effective form of birth control.
* Stable disease-modifying treatment for the last 2 months.
* Well controlled hypertension (stable antihypertensive medications for at least 2 months).
* BMI > 18 < 30.
* Written informed consent.

Exclusion Criteria:

* Exposure to a ketogenic diet or intermittent fasting for more than 2 weeks within 6 months before inclusion.

  * Significant weight-loss (> 10%) within 6 months before inclusion.
  * Diabetes mellitus.
  * Conditions prohibiting the use of a ketogenic diet (liver damage, pancreatic failure, pyruvate-carboxylase deficiency, defects in fatty acid oxidation/gluconeogenesis/ketolysis/neogenesis, hyperinsulinism), based on patient history.
  * Diagnosis with any disorder of fatty acid metabolism based on patient history.
  * Eating disorder.
  * Alcohol abuse.
  * Contraindication for MRI.
  * Participation in other interventional trial.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Observance | 56 days
  Objective observance (ketone body levels ≥0.8 mmol/l in ≥75% of blood measurements and ≥60% of maximal theoretic dose determined by used packages and self-report)
Feasibility | 56 days
  Patient reported feasibility, defined as a cohen d effect size of < 0.5 in the ADPKD impact scale.Both targets (observance and self-reported feasibility) must be met to reach the endpoint.

SECONDARY OUTCOMES:
Total Kidney Volume | 56 days
  Change in Total kidney volume (in mL; assessed with MRI) baseline vs day 56
Kidney Function | 56 days
  Change in estimated glomerular filtration rate (eGFR) according to CKD-EPI; baseline vs day 56

IPD SHARING:
Plan to Share IPD: Undecided